CLINICAL TRIAL: NCT04832945
Title: Multicenter Retrospective Cohort Study of Ivermectin as a SARS-CoV-2 Pre-exposure Prophylactic Method in Healthcare Workers in Dominican Republic
Brief Title: SARS-CoV-2 Pre-exposure Prophylaxis With Ivermectin Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Grupo Rescue S.A.S República Dominicana (Network)
Responsible Party: Sponsor
Other Study IDs: 8953
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Ivermectin; SARS-CoV-2; Coronavirus; Prophylaxis; PrEP; Covid-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Ivermectin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ivermectin Group: Healthcare personnel receiving Ivermectin weekly PrEP
  Interventions: Drug: Ivermectin 6 Mg Oral Tablet
- Control Group: Healthcare personnel not receiving Ivermectin

INTERVENTIONS:
Drug: Ivermectin 6 Mg Oral Tablet — Ivermectin weekly oral dose 0.2 mg/kg equivalent for 4 weeks
  Other Names: Ivermectin
  Groups: Ivermectin Group

SUMMARY:
This observational study, a multicenter retrospective cohort database study, carried out in two medical centers, Centro Medico Bournigal (CMBO) in Puerto Plata and Centro Medico Punta Cana (CMPC) in Punta Cana, Dominican Republic, sought to determine whether Ivermectin, at a weekly orally dose of 0.2 mg/kg, is an effective pre-exposure prophylactic method (PrEP) for the spread of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), in the healthcare workers. The study began on June 29, 2020 and ended on July 26, 2020 (4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Active workers from Centro Medico Bournigal (CMBO) and Centro Medico Punta Cana (CMPC) during the study.

Exclusion Criteria

* Workers with positive Covid-19 RT-PCR prior to the start of the study
* Those that did not take the first dose of Ivermectin the first week at the start of the study
* Those that did not complied with at least 2 out of 4 weekly doses
* Those that had greater than 14 days difference in days between two intakes Ivermectin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers who was part of Ivermectin prophylaxis program and signed the informed consent at CMPC and CMBO in Dominican Republic was analyzed and included in the intervention group. Those who didn't participate in the prophylaxis program but were on active duty during the 4 weeks of the study were included in the control group.
  Workers excluded from Ivermectin prophylaxis program was:
  * Pregnant or suspected pregnant women
  * Women breastfeeding
  * Patients receiving coumarin anticoagulants
  * Those allergic to Ivermectin
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants RT-PCR positive for Covid-19 | 4 weeks
  Workers confirmed Covid-19 through Reverse Transcription Polymerase Chain Reaction (RT-PCR) test

SECONDARY OUTCOMES:
Number of sick participants who condition deteriorated | 4 weeks
  Workers infected with Covid-19, confirmed with RT-PCR and required hospitalization and/or ICU
Number of sick participants who died | 4 weeks
  Workers infected with Covid-19, confirmed with RT-PCR and died.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Morgenstern, MD, Principal Investigator — Grupo Rescue; Jose Natalio Redondo, MD, Principal Investigator — Grupo Rescue; Alvaro Olavarria, Data Analyst, Principal Investigator — Grupo Rescue
Locations (2):
- Dominican Republic (2):
  - Centro Medico Bournigal, Puerto Plata
  - Centro Médico Punta Cana, Punta Cana

IPD SHARING:
Plan to Share IPD: No